CLINICAL TRIAL: NCT02698189
Title: A Phase IB Trial With MK-8628, a Small Molecule Inhibitor of the Bromodomain and Extra-Terminal (BET) Proteins, in Subjects With Selected Hematologic Malignancies
Brief Title: A Dose Exploration Study With Birabresib (MK-8628) in Participants With Selected Hematologic Malignancies (MK-8628-005)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated due to limited efficacy and not due to safety reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8628-005; MK-8628-005 (Other: Merck Protocol Number); 2015-005487-42 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-03 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: AML Including AML de Novo and AML Secondary to MDS; DLBCL
MeSH Terms: interventions — OTX015

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Birabresib 20 mg AML Cohort (Experimental): Participants in the AML cohort received 20 mg of birabresib as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
  Interventions: Drug: Birabresib Dose 20 mg
- Birabresib 20 mg DLBCL Cohort (Experimental): Participants in the DLBCL cohort received 20 mg of birabresib as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
  Interventions: Drug: Birabresib Dose 20 mg

INTERVENTIONS:
Drug: Birabresib Dose 20 mg — Administered as an oral capsule twice a day for 21 consecutive days per cycle.
  Other Names: OTX015; MK-8628

SUMMARY:
This is a study to determine the recommended dose of birabresib (MK-8628) for further studies in participants with acute myeloid leukemia (AML) including AML de novo and AML secondary to myelodysplastic syndrome (MDS) and in participants with diffuse large B cell lymphoma (DLBCL). The recommended dose will be established by evaluating dose limiting toxicity (DLT), safety, tolerability, and early efficacy signals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML (AML de novo and post-MDS) or DLBCL
* AML participants must have the following malignancy criteria: measurable and evaluable disease per tumor response criteria; ≥ 5% bone marrow blasts without alternate causality; and > 90 days since allogeneic stem cell transplantation relapse in participants relapsing after transplant
* AML participants who are Philadelphia chromosome positive must have received ≥ 2 lines of therapy, including 2 bcr-abl tyrosine-kinase (TK) inhibitors (among imatinib, nilotinib and dasatinib), or only 1 line including 1 TK inhibitor if the relapse/refractoriness is associated with the detection of a resistance mutation to these inhibitors
* AML participants < 60 years old must be in second or further relapse or relapsing after allogeneic stem cell transplantation regardless of number of relapses
* AML participants ≥ 60 years old in first relapse with a disease-free interval < 12 months, or further relapse. First relapse is also applicable to AML post-MDS patients who have received prior treatment for MDS, but have not received prior treatment for AML.
* DLBCL participants must have the following malignancy criteria: measurable and evaluable disease per tumor response criteria and ≥ 1 tumor mass that is ≥ 15 mm (long axis of lymph node) or ≥ 10 mm (short axis of lymph node or extranodal lesions) on spiral CT scan; failed 2 standard lines of therapy (at least one containing an anti-CD20 monoclonal antibody), or for whom such treatment is contraindicated.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1
* An interval of ≥3 weeks since chemotherapy (≥ 6 weeks for nitrosoureas or mitomycin C), immunotherapy, hormone therapy or any other anticancer therapy or surgical intervention resection, or ≥3 half-lives for monoclonal antibodies, or ≥ 5 half-lives for other non-cytotoxic agents (whichever is longer)
* Female participants must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours of study start)
* Female and male participants of reproductive potential must agree to use adequate contraception starting from the first dose of trial treatment through 90 days after the last dose of study medication

Exclusion Criteria:

* Known primary central nervous system (CNS) malignancy or symptomatic or untreated CNS metastases
* History of prior or concomitant malignancies within 3 years of study start
* Has other serious illness or medical condition, such as active infection, unresolved bowel obstruction, psychiatric disorders, or cerebrovascular accident within 1 year of study start
* Known history of human immunodeficiency virus (HIV) and/or active Hepatitis B or C infections
* Has one of the following cardiac-related conditions: Congestive heart failure; angina pectoris; myocardial infarction (within 1 year of study start); uncontrolled hypertension; or uncontrolled arrhythmias
* Is receiving other concomitant anticancer treatment
* Has received high dose chemotherapy followed by autologous stem cell transplantation less than 90 days prior to first dose of study treatment
* Is receiving concomitant therapy with strong CYP3A4 or CYP2A6 inhibitors or inducers
* Is pregnant or breast-feeding
* Participation in a clinical trial involving an investigational drug within 30 days of study start
* Known additional malignancy that is progressing or requires active treatment
* Has been previously treated with a Bromodomain and Extra-terminal (BET) inhibitor
* Has acute promyelocytic leukemia, clinically uncontrolled disseminated intravascular coagulation, or peripheral cytopenia
* Has chronic graft versus host disease (GVHD) or on immunosuppressive therapy for the control of GVHD
* Has uncontrolled disease-related metabolic disorder
* Unable to swallow oral medications, or has gastrointestinal condition deemed to jeopardize intestinal absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment to the study was discontinued early based on a decision to terminate the MK-8628 program and based on limited efficacy signals and not due to safety-related concerns.
Groups:
- MK-8628 20 mg Acute Myeloid Leukemia (AML) Cohort: Participants in the AML cohort received 20 mg of MK-8628 as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
- MK-8628 20 mg Diffuse Large B Cell Lymphoma (DLBCL) Cohort: Participants in the DLBCL cohort received 20 mg of MK-8628 as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
Period: Overall Study
Arm/Group | MK-8628 20 mg Acute Myeloid Leukemia (AML) Cohort | MK-8628 20 mg Diffuse Large B Cell Lymphoma (DLBCL) Cohort
Started | 3 | 6
Completed | 0 | 0
Not Completed | 3 | 6
Not completed — Physician Decision | 3 | 0
Not completed — Progressive disease | 0 | 5
Not completed — Study terminated by sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- MK-8628 20 mg AML Cohort: Participants in the AML cohort received 20 mg of MK-8628 as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
- MK-8628 20 mg DLBCL Cohort: Participants in the DLBCL cohort received 20 mg of MK-8628 as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
- Total: Total of all reporting groups
Arm/Group | MK-8628 20 mg AML Cohort | MK-8628 20 mg DLBCL Cohort | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (17.3) | 63.8 (17.8) | 60.6 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Log2 Transformed Normalized Gene Expression Ratios (GERs) [Mean (Standard Deviation); unit: Gene expression ratio (Log2 scale)] — GERs for 49 Bromodomain and Extra-Terminal (BET) target genes were measured using messenger Ribonucleic Acid (mRNA) predose on Day 1 of Cycle 1 (21-day cycle). The expression level of target genes was quantitated by quantitative polymerase chain reaction and the data were normalized by the delta-delta cycle threshold (Ct) method using housekeeping genes. Baseline normalized GERs were expressed in logarithmic scale with a base of 2 (Log2 scale). Positive values=greater expression and negative values=reduced expression of any gene relative to housekeeping genes.
  Gene expression ratio (Log2 scale)
    Agmatinase (AGMAT) | -4.659 (0.888) | -3.731 (0.573) | -4.040 (0.786)
    Annexin A3 (ANXA3) | -2.568 (1.944) | 0.602 (1.399) | -0.455 (2.163)
    Atonal BHLH Transcription Factor 8 (ATOH8) | -6.560 (0.756) | -4.511 (0.851) | -5.194 (1.283)
    B-cell Lymphoma Extra Large (BCL.xL) | 2.744 (1.893) | 5.704 (1.588) | 4.718 (2.159)
    B-cell Lymphoma 2 (BCL2) | 0.699 (1.369) | 0.479 (0.979) | 0.552 (1.039)
    Bone Marrow X-linked Kinase (BMX) | -6.109 (0.357) | -2.408 (1.113) | -3.642 (2.057)
    Caspase Recruitment Domain Family Member 6 (CARD6) | -1.604 (0.490) | -1.074 (0.364) | -1.251 (0.462)
    C-C Motif Chemokine Receptor 1 (CCR1) | -1.566 (1.720) | 1.405 (0.863) | 0.415 (1.847)
    Cluster of Differentiation 163 (CD163) | -4.586 (1.591) | -1.789 (0.975) | -2.722 (1.784)
    Choline Kinase Alpha (CHKA) | 1.255 (0.670) | -0.795 (0.453) | -0.112 (1.136)
    Chemerin Chemokine-Like Receptor 1 (CMKLR1) | -1.967 (0.997) | -0.952 (1.111) | -1.290 (1.130)
    Cysteine/Serine-Rich Nuclear Protein 2 (CSRNP2) | -2.934 (0.399) | -2.765 (0.228) | -2.821 (0.282)
    Dicarbonyl and L-xylulose Reductase (DCXR) | 0.026 (0.230) | -0.326 (0.121) | -0.209 (0.231)
    Deoxyribonuclease 1 Like 3 (DNASE1L3) | -5.842 (1.960) | -4.857 (1.411) | -5.186 (1.564)
    Fc Gamma Receptor Ia (FCGR1A) | -2.119 (2.707) | 1.992 (1.363) | 0.622 (2.687)
    Fibroblast Growth Factor Receptor 1 (FGFR1) | -3.202 (2.427) | -3.761 (0.669) | -3.574 (1.353)
    G Protein-Coupled Receptor 141 (GPR141) | -2.185 (0.603) | -2.022 (0.511) | -2.076 (0.511)
    Granzyme A (GZMA) | -0.640 (2.151) | 2.416 (1.002) | 1.397 (2.029)
    Granzyme B (GZMB) | -0.175 (3.390) | 2.558 (1.025) | 1.647 (2.323)
    Granzyme K (GZMK) | -1.730 (2.427) | 0.576 (1.356) | -0.193 (1.988)
    H2A Histone Family Member X (H2AFX) | -0.504 (0.215) | -1.629 (0.379) | -1.254 (0.646)
    Hepatitis A Virus Cellular Receptor 2 (HAVCR2) | -1.177 (0.391) | -0.210 (0.670) | -0.532 (0.744)
    Class B Basic Helix-Loop-Helix Protein 41 (HES6) | -4.202 (1.520) | -3.679 (1.156) | -3.853 (1.217)
    Hexamethylene Bisacetamide Inducible 1 (HEXIM1) | 0.037 (0.788) | 0.803 (0.229) | 0.548 (0.579)
    Hepatocyte Growth Factor (HGF) | 1.880 (3.142) | -0.798 (0.668) | 0.095 (2.131)
    Histone Cluster 2 H2B Family Member F (HIST2H2BF) | 2.317 (2.412) | 3.848 (0.440) | 3.337 (1.470)
    Inhibitor of Nuclear Factor-kB (IKBKE) | -0.358 (0.494) | -0.019 (0.186) | -0.132 (0.334)
    Interleukin 12 Receptor Subunit Beta 2 (IL12RB2) | -3.576 (2.016) | -2.592 (1.437) | -2.920 (1.596)
    Interleukin 7 Receptor (IL7R) | -0.531 (2.292) | 2.816 (0.829) | 1.700 (2.131)
    Lunatic Fringe (Drosophila) Homolog (LFNG) | -0.931 (0.722) | 0.671 (0.549) | 0.137 (0.980)
    Leukocyte Immunoglobulin Like Receptor A4 (LILRA4) | -6.838 (1.271) | -3.803 (1.630) | -4.815 (2.090)
    Macrophage Receptor (MARCO) | -5.927 (0.816) | -1.022 (1.370) | -2.657 (2.712)
    Membrane Spanning 4-Domains A2 (MS4A2) | -3.308 (2.486) | -4.689 (1.515) | -4.229 (1.859)
    Class E Basic Helix-Loop-Helix Protein 39 (MYC) | 1.727 (0.155) | -0.004 (0.739) | 0.573 (1.047)
    Nudix Hydrolase 12 (NUDT12) | -3.948 (2.918) | -4.204 (0.700) | -4.118 (1.566)
    Proliferating Cell Nuclear Antigen (PCNA) | -0.861 (0.241) | -2.212 (0.484) | -1.762 (0.786)
    Protein Tyrosine Phosphatase PTP-U2 (PTPRO) | -4.546 (1.000) | -2.704 (0.426) | -3.318 (1.101)
    C17orf87 (SCIMP) | -3.588 (2.237) | 1.073 (0.589) | -0.481 (2.626)
    Serpin Family G Member 1 (SERPING1) | 0.208 (1.584) | 0.864 (1.168) | 0.645 (1.260)
    CD353 Antigen (SLAMF8) | -3.950 (1.981) | -2.729 (0.847) | -3.136 (1.342)
    Stathmin 1 (STMN1) | 2.382 (0.359) | -0.358 (0.828) | 0.556 (1.529)
    Thyroglobulin (TG) | -4.955 (1.255) | -4.221 (0.440) | -4.465 (0.806)
    TIFA Inhibitor (TIFAB) | -2.808 (1.959) | -2.905 (0.754) | -2.873 (1.148)
    Transmembrane Protein 150B (TMEM150B) | -5.664 (0.887) | -2.105 (0.391) | -3.291 (1.859)
    Lymphocyte Activation Antigen CD30 (TNFRSF8) | -4.865 (0.886) | -0.925 (0.938) | -2.238 (2.151)
    B-Cell-Activating Factor (TNFSF13B) | 0.117 (1.746) | 1.595 (0.587) | 1.103 (1.235)
    Tuftelin 1 (TUFT1) | -6.288 (1.491) | -4.377 (0.519) | -5.014 (1.280)
    Nemitin (WDR47) | -1.748 (0.319) | -1.377 (0.139) | -1.501 (0.268)
    X-C Motif Chemokine Ligand 2 (XCL2) | -2.728 (0.852) | -0.820 (1.313) | -1.456 (1.473)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Dose Limiting Toxicity (DLT)
Description: DLT was any of the following drug related (DR) investigator-assessed adverse events: pancytopenia with hypocellular bone marrow and no marrow blasts lasting for ≥6 weeks; Grade (G)4 hematologic toxicity lasting ≥7 days except thrombocytopenia; G4 thrombocytopenia; G3 thrombocytopenia with bleeding; G3 or 4 febrile or infection-related neutropenia; G4 nonhematologic (NH) toxicity (not laboratory); G3 NH toxicity (not laboratory), nausea, vomiting, or diarrhea lasting >3 days despite supportive care; G3 or 4 NH laboratory abnormality requiring medical intervention, hospitalization, or persisting >1 week; increases in alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin, or international normalization ratio indicative of significant liver impairment; DR adverse event leading to discontinuation or ≥20% missed planned doses in Cycle 1; DR toxicity causing >2 week delay in starting Cycle 2; or G5 toxicity.
Time Frame: From time of first dose up to the end of Cycle 1 (21-day cycle): up to 21 days
Population: The population consisted of all participants that received at least 85% of the planned dose of study drug (18 days) or experienced a DLT during Cycle 1 (21-day cycle).
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8628 20 mg AML Cohort | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 2 | 6
Percentage of participants | 0.00 | 16.67
Statistical Analysis 1: Comparison: MK-8628 20 mg AML Cohort; Test type: Other — 80% Bayesian credible interval based on a prior distribution of Beta (1, 1); 80% 2-sided Bayesian credible interval: lower = 0.000; upper = 0.415
Statistical Analysis 2: Comparison: MK-8628 20 mg DLBCL Cohort; Test type: Other — 80% Bayesian credible interval based on a prior distribution of Beta (1, 1); 80% 2-sided Bayesian credible interval: lower = 0.040; upper = 0.391

2. Secondary Outcome: Percentage of Participants Who Experienced At Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of all participants who experienced at least one AE is presented. Per protocol, these results are based on a data cutoff date of 09-May-2018.
Time Frame: From time of first dose until the end of follow-up (up to 8 months)
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8628 20 mg AML Cohort | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 3 | 6
Percentage of participants | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The percentage of all participants who discontinued study treatment due to an AE is presented. Per protocol, these results are based on a data cutoff date of 09-May-2018.
Time Frame: From time of first dose until the end of treatment (up to 7 months)
Population: The analysis population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | MK-8628 20 mg AML Cohort | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 3 | 6
Percentage of participants | 0.0 | 0.0

4. Secondary Outcome: Objective Response Rate (ORR) in the Acute Myeloid Leukemia (AML) Cohort Per International Working Group Criteria: European LeukemiaNet (Döhner et al, Blood, 2010)
Description: ORR was defined as the percentage of the participants who had complete response (CR) or partial response (PR) as assessed by investigator review. Participants in the AML cohort were assessed using bone marrow aspiration and hematologic criteria and response was evaluated based on European LeukemiaNet (Döhner et al, Blood, 2010). The criteria for complete response included: bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 × 10^9/Liter; platelet count >100 × 10^9/Liter; and independence of red cell transfusions. The criteria for partial response included: decrease of bone marrow blast percentage to 5% to 25%; decrease of pretreatment bone marrow blast percentage by at least 50%; and all hematologic criteria associated with CR. The percentage of participants who achieved CR or PR is presented.
Time Frame: Every 3 weeks starting from Cycle 2 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the AML cohort who received at least one dose of study treatment and had data evaluable for ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-8628 20 mg AML Cohort
Number analyzed (Participants) | 3
Percentage of participants
  Complete response | 0.0 [0.0 to 70.8]
  Partial response | 0.0 [0.0 to 70.8]

5. Secondary Outcome: Objective Response Rate (ORR) in the Diffuse Large B Cell Lymphoma (DLBCL) Cohort Per International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014)
Description: ORR was defined as the percentage of the participants who had complete response (CR) or partial response (PR) as assessed by investigator review. Participants in the DLBCL cohort were assessed using computed tomography (CT) and positron emission tomography (PET)-CT and response was evaluated based on the Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). The criteria for CR included complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. The criteria for PR included: partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants who achieved CR or PR is presented.
Time Frame: Every 12 weeks starting from Cycle 5 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the DLBCL cohort who received at least one dose of study treatment and had data evaluable for ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 6
Percentage of participants
  Complete response | 0.0 [0.0 to 45.9]
  Partial response | 16.7 [0.4 to 64.1]

6. Secondary Outcome: Duration of Response (DOR) in the Acute Myeloid Leukemia (AML) Cohort Per International Working Group Criteria: European LeukemiaNet (Döhner et al, Blood, 2010)
Description: DOR was defined as the time from complete response (CR) or partial response (PR) to documented disease progression or death as assessed by investigator review. Participants in the AML cohort were assessed using bone marrow aspiration and hematologic criteria and response was evaluated based on European LeukemiaNet (Döhner et al, Blood, 2010). The criteria for complete response included: bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 × 10^9/Liter; platelet count >100 × 10^9/Liter; and independence of red cell transfusions. The criteria for partial response included: decrease of bone marrow blast percentage to 5% to 25%; decrease of pretreatment bone marrow blast percentage by at least 50%; and all hematologic criteria associated with CR.
Time Frame: Every 3 weeks starting from Cycle 2 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the AML cohort who received at least one dose of study treatment and had data evaluable for DOR analysis. DOR could not be calculated because no participants met criteria for analysis: CR or PR and documented disease progression or death.
Arm/Group | MK-8628 20 mg AML Cohort
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Response (DOR) in the Diffuse Large B Cell Lymphoma (DLBCL) Cohort Per International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014)
Description: DOR was defined as the time from complete response (CR) or partial response (PR) to documented disease progression or death as assessed by investigator review. Participants in the DLBCL cohort were assessed using computed tomography (CT) and positron emission tomography (PET)-CT and response was evaluated based on the Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). The criteria for CR included complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. The criteria for PR included: partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal).
Time Frame: Every 12 weeks starting from Cycle 5 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the DLBCL cohort who received at least one dose of study treatment and had data evaluable for DOR analysis. DOR could not be calculated because no participants met criteria for analysis: CR or PR and documented disease progression or death.
Arm/Group | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 0

8. Secondary Outcome: Disease Control Rate (DCR) in the Acute Myeloid Leukemia (AML) Cohort Per International Working Group Criteria: European LeukemiaNet (Döhner et al, Blood, 2010)
Description: DCR was defined as the percentage of the participants who had stable disease, complete response (CR) or partial response (PR) as assessed by investigator review. Participants in the AML cohort were assessed using bone marrow aspiration and hematologic criteria and response was evaluated based on European LeukemiaNet (Döhner et al, Blood, 2010). The criteria for complete response included: bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 × 10^9/Liter; platelet count >100 × 10^9/Liter; and independence of red cell transfusions. The criteria for partial response included: decrease of bone marrow blast percentage to 5% to 25%; decrease of pretreatment bone marrow blast percentage by at least 50%; and all hematologic criteria associated with CR.
Time Frame: Every 3 weeks starting from Cycle 2 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the AML cohort who received at least one dose of study treatment and had data evaluable for DCR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-8628 20 mg AML Cohort
Number analyzed (Participants) | 3
Percentage of participants
  Complete response | 0.0 [0.0 to 70.8]
  Partial response | 0.0 [0.0 to 70.8]
  Stable disease | 0.0 [0.0 to 70.8]

9. Secondary Outcome: Disease Control Rate (DCR) in the Diffuse Large B Cell Lymphoma (DLBCL) Cohort Per International Working Group Criteria: Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014)
Description: DCR was defined as the percentage of the participants in the DLBCL cohort who had stable disease, complete response (CR) or partial response (PR) as assessed by investigator review. Participants in the DLBCL cohort were assessed using computed tomography (CT) and positron emission tomography (PET)-CT and response was evaluated based on the Lugano Classification (Cheson et al, Journal of Clinical Oncology, 2014). The criteria for CR included complete metabolic (no/minimal fluorodeoxyglucose [FDG] uptake) and radiologic response (target lesions regress to ≤5 cm in longest transverse diameter of a lesion) and no new lesions. The criteria for PR included: partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of the product of the perpendicular diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal).
Time Frame: Every 12 weeks starting from Cycle 5 (21-day cycle) until disease progression (up to 7 months)
Population: The analysis population consisted of all participants in the DLBCL cohort who received at least one dose of study treatment and had data evaluable for DCR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MK-8628 20 mg DLBCL Cohort
Number analyzed (Participants) | 6
Percentage of participants
  Complete response | 0.0 [0.0 to 45.9]
  Partial response | 16.7 [0.4 to 64.1]
  Stable disease | 0.0 [0.0 to 45.9]

10. Secondary Outcome: Observed Maximum Concentration (Cmax) of MK-8628
Description: Blood samples were collected to determine Cmax at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, Cmax for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The Cmax of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for Cmax analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MK-8628 20 mg AML+DLBCL Cohorts: Total number of participants from both cohorts (AML and DLBCL) received 20 mg of MK-8628 as an oral capsule twice a day for 21 consecutive days per cycle (21-day cycle).
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 9
ng/mL | 360 (132)

11. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8628
Description: Blood samples were collected to determine Tmax at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, Tmax for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The Tmax of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for the Tmax analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 9
hr | 2.25 [1.00 to 8.00]

12. Secondary Outcome: Observed Minimum Concentration (Cmin) of MK-8628
Description: Blood samples were collected to determine Cmin at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, Cmin for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The Cmin of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for the Cmin analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 9
ng/mL | 134 (77.2)

13. Secondary Outcome: Area Under the Concentration-Time Curve of MK-8628 From Time 0 to Infinity (AUC 0-∞)
Description: Blood samples were collected to determine AUC 0-∞ at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, AUC 0-∞ for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The AUC 0-∞ of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for the AUC 0-∞ analysis.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
hr*ng/mL | 3580 (1340)

14. Secondary Outcome: Apparent Terminal Half-life (t1/2) for MK-8628
Description: Blood samples were collected to determine t1/2 at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, t1/2 for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The t1/2 of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for the t1/2 analysis.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
hr | 7.62 (2.94)

15. Secondary Outcome: Apparent Total Body Clearance (CL/F) of MK-8628
Description: Blood samples were collected to determine CL/F at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, CL/F for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The CL/F of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for CL/F analysis.
Measure: Mean (Standard Deviation); unit: Liters/hr
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
Liters/hr | 6.46 (2.70)

16. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of MK-8628
Description: Blood samples were collected to determine Vz/F at the following time points: Cycle 1 (21-day cycle) Day 1 at predose and 20 minutes, 1 hour, 2.25 hours, 3.25 hours, 8 hours and 12 hours postdose; Cycle 1 (21-day cycle) at predose on Days 8 and 15; and Cycle 2 (21-day cycle) at predose on Day 1. Per protocol, Vz/F for MK-8628 was assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The Vz/F of MK-8628 after oral administration is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose.
Time Frame: Up to 22 days post MK-8628 dose
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received at least one dose of MK-8628 20 mg and had data available for Vz/F analysis.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
Liters | 65.6 (24.3)

17. Secondary Outcome: Change From Baseline in Bromodomain and Extra-Terminal Domain (BET) Protein Target Gene Expression at 3 Hours Postdose on Day 1 of Cycle 1 (21-day Cycle)
Description: Fold change from baseline (predose on Day 1 of Cycle 1 [21-day cycle]) in normalized gene expression ratios (nGER) for 49 target genes was measured to assess target engagement of BET proteins predose and 3 hours postdose using quantitative polymerase chain reaction (qPCR). Data were normalized by the delta-delta cycle threshold (Ct) method using housekeeping genes. Fold change from baseline was calculated as nGER at 3 hours postdose Day 1/baseline in logarithmic scale with a base of 2 (Log2 scale). Per protocol, target genes were assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The fold change in nGER for each target gene is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose. A two-fold increase in gene expression indicated a +1 Log2 fold change. Conversely, a two-fold decrease in gene expression indicated a -1 Log2 fold change.
Time Frame: Baseline (predose on Day 1 of Cycle 1 [21-day cycle]) and 3 hours postdose on Day 1 of Cycle 1 (21-day cycle)
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received one dose of MK-8628 20 mg on Day 1 of Cycle 1 (21-day cycle) and had data available for the gene expression analysis.
Measure: Mean (Standard Deviation); unit: Log2 scale fold change
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 9
Log2 scale fold change
  Agmatinase (AGMAT) | -0.466 (0.266)
  Annexin A3 (ANXA3) | -0.182 (0.537)
  Atonal BHLH Transcription Factor 8 (ATOH8) | -0.296 (0.627)
  B-cell Lymphoma Extra Large (BCL.xL) | -0.219 (0.791)
  B-cell Lymphoma 2 (BCL2) | -0.053 (0.289)
  Bone Marrow X-linked Kinase (BMX) | -0.093 (0.718)
  Caspase Recruitment Domain Family Member 6 (CARD6) | -0.245 (0.371)
  C-C Motif Chemokine Receptor 1 (CCR1) | -0.246 (0.351)
  Cluster of Differentiation 163 (CD163) | -0.457 (0.594)
  Choline Kinase Alpha (CHKA) | 0.110 (0.309)
  Chemerin Chemokine-Like Receptor 1 (CMKLR1) | -0.194 (0.465)
  Cysteine/Serine-Rich Nuclear Protein 2 (CSRNP2) | 0.150 (0.190)
  Dicarbonyl and L-xylulose Reductase (DCXR) | 0.300 (0.211)
  Deoxyribonuclease 1 Like 3 (DNASE1L3) | -0.305 (0.614)
  Fc Gamma Receptor Ia (FCGR1A) | -0.360 (0.483)
  Fibroblast Growth Factor Receptor 1 (FGFR1) | 0.127 (0.382)
  G Protein-Coupled Receptor 141 (GPR141) | 0.054 (0.546)
  Granzyme A (GZMA) | -0.198 (0.768)
  Granzyme B (GZMB) | -0.163 (0.262)
  Granzyme K (GZMK) | -0.127 (0.602)
  H2A Histone Family Member X (H2AFX) | 0.049 (0.161)
  Hepatitis A Virus Cellular Receptor 2 (HAVCR2) | -0.272 (0.172)
  Class B Basic Helix-Loop-Helix Protein 41 (HES6) | 0.189 (0.594)
  Hexamethylene Bisacetamide Inducible 1 (HEXIM1) | 0.315 (0.234)
  Hepatocyte Growth Factor (HGF) | -0.461 (0.234)
  Histone Cluster 2 H2B Family Member F (HIST2H2BF) | 0.325 (0.346)
  Inhibitor of Nuclear Factor-kB (IKBKE) | -0.124 (0.243)
  Interleukin 12 Receptor Subunit Beta 2 (IL12RB2) | 0.012 (0.334)
  Interleukin 7 Receptor (IL7R) | 0.003 (0.470)
  Lunatic Fringe (Drosophila) Homolog (LFNG) | 0.182 (0.188)
  Leukocyte Immunoglobulin Like Receptor A4 (LILRA4) | -0.403 (0.590)
  Macrophage Receptor (MARCO) | -0.321 (0.417)
  Membrane Spanning 4-Domains A2 (MS4A2) | -0.646 (0.850)
  Class E Basic Helix-Loop-Helix Protein 39 (MYC) | -0.359 (0.406)
  Nudix Hydrolase 12 (NUDT12) | -0.309 (0.671)
  Proliferating Cell Nuclear Antigen (PCNA) | 0.093 (0.270)
  Protein Tyrosine Phosphatase PTP-U2 (PTPRO) | -0.391 (0.488)
  C17orf87 (SCIMP) | -0.159 (0.328)
  Serpin Family G Member 1 (SERPING1) | -0.137 (0.579)
  CD353 Antigen (SLAMF8) | -0.485 (0.434)
  Stathmin 1 (STMN1) | -0.054 (0.199)
  Thyroglobulin (TG) | 0.485 (0.377)
  TIFA Inhibitor (TIFAB) | -0.405 (0.334)
  Transmembrane Protein 150B (TMEM150B) | -0.283 (0.482)
  Lymphocyte Activation Antigen CD30 (TNFRSF8) | -0.522 (0.312)
  B-Cell-Activating Factor (TNFSF13B) | -0.135 (0.299)
  Tuftelin 1 (TUFT1) | 0.282 (0.544)
  Nemitin (WDR47) | 0.144 (0.162)
  X-C Motif Chemokine Ligand 2 (XCL2) | -0.365 (0.419)

18. Secondary Outcome: Change From Baseline in Bromodomain and Extra-Terminal Domain (BET) Protein Target Gene Expression at 8 Hours Postdose on Day 1 of Cycle 1 (21-day Cycle)
Description: Fold change from baseline (predose on Day 1 of Cycle 1 [21-day cycle]) in normalized gene expression ratios (nGER) for 49 target genes was measured to assess target engagement of BET proteins predose and 8 hours postdose using quantitative polymerase chain reaction (qPCR). Data were normalized by the delta-delta cycle threshold (Ct) method using housekeeping genes. Fold change from baseline was calculated as nGER at 8 hours postdose Day 1/baseline in logarithmic scale with a base of 2 (Log2 scale). Per protocol, target genes were assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The fold change in nGER for each target gene is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose. A two-fold increase in gene expression indicated a +1 Log2 fold change. Conversely, a two-fold decrease in gene expression indicated a -1 Log2 fold change.
Time Frame: Baseline (predose on Day 1 of Cycle 1 [21-day cycle]) and 8 hours postdose on Day 1 of Cycle 1 (21-day cycle)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Log2 scale fold change
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
Log2 scale fold change
  Agmatinase (AGMAT) | -0.493 (0.322)
  Annexin A3 (ANXA3) | 0.111 (0.865)
  Atonal BHLH Transcription Factor 8 (ATOH8) | -0.049 (0.923)
  B-cell Lymphoma Extra Large (BCL.xL) | -0.169 (0.603)
  B-cell Lymphoma 2 (BCL2) | -0.133 (0.266)
  Bone Marrow X-linked Kinase (BMX) | -0.008 (1.008)
  Caspase Recruitment Domain Family Member 6 (CARD6) | -0.091 (0.324)
  C-C Motif Chemokine Receptor 1 (CCR1) | -0.257 (0.467)
  Cluster of Differentiation 163 (CD163) | -0.640 (0.994)
  Choline Kinase Alpha (CHKA) | -0.116 (0.384)
  Chemerin Chemokine-Like Receptor 1 (CMKLR1) | -0.218 (0.736)
  Cysteine/Serine-Rich Nuclear Protein 2 (CSRNP2) | 0.152 (0.350)
  Dicarbonyl and L-xylulose Reductase (DCXR) | 0.536 (0.187)
  Deoxyribonuclease 1 Like 3 (DNASE1L3) | -0.306 (0.661)
  Fc Gamma Receptor Ia (FCGR1A) | -0.126 (0.390)
  Fibroblast Growth Factor Receptor 1 (FGFR1) | 0.125 (0.295)
  G Protein-Coupled Receptor 141 (GPR141) | -0.085 (0.597)
  Granzyme A (GZMA) | -0.015 (1.103)
  Granzyme B (GZMB) | -0.262 (0.382)
  Granzyme K (GZMK) | 0.001 (0.898)
  H2A Histone Family Member X (H2AFX) | 0.082 (0.156)
  Hepatitis A Virus Cellular Receptor 2 (HAVCR2) | -0.294 (0.276)
  Class B Basic Helix-Loop-Helix Protein 41 (HES6) | 0.378 (0.888)
  Hexamethylene Bisacetamide Inducible 1 (HEXIM1) | 0.345 (0.234)
  Hepatocyte Growth Factor (HGF) | -0.325 (0.228)
  Histone Cluster 2 H2B Family Member F (HIST2H2BF) | 0.239 (0.372)
  Inhibitor of Nuclear Factor-kB (IKBKE) | -0.153 (0.262)
  Interleukin 12 Receptor Subunit Beta 2 (IL12RB2) | -0.018 (0.352)
  Interleukin 7 Receptor (IL7R) | 0.016 (0.461)
  Lunatic Fringe (Drosophila) Homolog (LFNG) | 0.104 (0.228)
  Leukocyte Immunoglobulin Like Receptor A4 (LILRA4) | -0.151 (0.494)
  Macrophage Receptor (MARCO) | -0.441 (0.777)
  Membrane Spanning 4-Domains A2 (MS4A2) | -0.232 (0.786)
  Class E Basic Helix-Loop-Helix Protein 39 (MYC) | -0.481 (0.611)
  Nudix Hydrolase 12 (NUDT12) | -0.295 (0.587)
  Proliferating Cell Nuclear Antigen (PCNA) | 0.036 (0.318)
  Protein Tyrosine Phosphatase PTP-U2 (PTPRO) | 0.037 (0.632)
  C17orf87 (SCIMP) | -0.246 (0.425)
  Serpin Family G Member 1 (SERPING1) | -0.162 (0.922)
  CD353 Antigen (SLAMF8) | -0.307 (0.297)
  Stathmin 1 (STMN1) | -0.091 (0.292)
  Thyroglobulin (TG) | 0.347 (0.724)
  TIFA Inhibitor (TIFAB) | -0.257 (0.586)
  Transmembrane Protein 150B (TMEM150B) | -0.136 (0.488)
  Lymphocyte Activation Antigen CD30 (TNFRSF8) | -0.830 (0.692)
  B-Cell-Activating Factor (TNFSF13B) | -0.112 (0.308)
  Tuftelin 1 (TUFT1) | 0.341 (0.546)
  Nemitin (WDR47) | 0.164 (0.243)
  X-C Motif Chemokine Ligand 2 (XCL2) | -0.190 (0.607)

19. Secondary Outcome: Change From Baseline in Bromodomain and Extra-Terminal Domain (BET) Protein Target Gene Expression at 12 Hours Postdose on Day 1 of Cycle 1 (21-day Cycle)
Description: Fold change from baseline (predose on Day 1 of Cycle 1 [21-day cycle]) in normalized gene expression ratios (nGER) for 49 target genes was measured to assess target engagement of BET proteins predose and 12 hours postdose using quantitative polymerase chain reaction (qPCR). Data were normalized by the delta-delta cycle threshold (Ct) method using housekeeping genes. Fold change from baseline was calculated as nGER at 12 hours postdose Day 1/baseline in logarithmic scale with a base of 2 (Log2 scale). Per protocol, target genes were assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The fold change in nGER for each target gene is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose. A two-fold increase in gene expression indicated a +1 Log2 fold change. Conversely, a two-fold decrease in gene expression indicated a -1 Log2 fold change.
Time Frame: Baseline (predose on Day 1 of Cycle 1 [21-day cycle]) and 12 hours postdose on Day 1 of Cycle 1 (21-day cycle)
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received two doses of MK-8628 20 mg on Day 1 of Cycle 1 (21-day cycle) and had data available for the gene expression analysis.
Measure: Mean (Standard Deviation); unit: Log2 scale fold change
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
Log2 scale fold change
  Agmatinase (AGMAT) | -0.287 (0.248)
  Annexin A3 (ANXA3) | 0.020 (0.863)
  Atonal BHLH Transcription Factor 8 (ATOH8) | -0.363 (0.649)
  B-cell Lymphoma Extra Large (BCL.xL) | -0.071 (0.500)
  B-cell Lymphoma 2 (BCL2) | -0.078 (0.313)
  Bone Marrow X-linked Kinase (BMX) | 0.047 (0.781)
  Caspase Recruitment Domain Family Member 6 (CARD6) | -0.052 (0.241)
  C-C Motif Chemokine Receptor 1 (CCR1) | -0.108 (0.380)
  Cluster of Differentiation 163 (CD163) | -0.528 (0.734)
  Choline Kinase Alpha (CHKA) | -0.191 (0.343)
  Chemerin Chemokine-Like Receptor 1 (CMKLR1) | -0.078 (0.510)
  Cysteine/Serine-Rich Nuclear Protein 2 (CSRNP2) | 0.128 (0.328)
  Dicarbonyl and L-xylulose Reductase (DCXR) | 0.511 (0.379)
  Deoxyribonuclease 1 Like 3 (DNASE1L3) | -0.074 (0.409)
  Fc Gamma Receptor Ia (FCGR1A) | -0.126 (0.534)
  Fibroblast Growth Factor Receptor 1 (FGFR1) | 0.193 (0.304)
  G Protein-Coupled Receptor 141 (GPR141) | 0.040 (0.673)
  Granzyme A (GZMA) | -0.110 (0.841)
  Granzyme B (GZMB) | -0.225 (0.370)
  Granzyme K (GZMK) | -0.034 (0.648)
  H2A Histone Family Member X (H2AFX) | -0.013 (0.169)
  Hepatitis A Virus Cellular Receptor 2 (HAVCR2) | -0.181 (0.239)
  Class B Basic Helix-Loop-Helix Protein 41 (HES6) | 0.257 (0.654)
  Hexamethylene Bisacetamide Inducible 1 (HEXIM1) | 0.308 (0.260)
  Hepatocyte Growth Factor (HGF) | -0.298 (0.241)
  Histone Cluster 2 H2B Family Member F (HIST2H2BF) | 0.288 (0.451)
  Inhibitor of Nuclear Factor-kB (IKBKE) | -0.092 (0.224)
  Interleukin 12 Receptor Subunit Beta 2 (IL12RB2) | 0.035 (0.466)
  Interleukin 7 Receptor (IL7R) | 0.051 (0.316)
  Lunatic Fringe (Drosophila) Homolog (LFNG) | 0.167 (0.202)
  Leukocyte Immunoglobulin Like Receptor A4 (LILRA4) | -0.023 (0.396)
  Macrophage Receptor (MARCO) | -0.714 (0.507)
  Membrane Spanning 4-Domains A2 (MS4A2) | -0.332 (0.658)
  Class E Basic Helix-Loop-Helix Protein 39 (MYC) | -0.376 (0.528)
  Nudix Hydrolase 12 (NUDT12) | -0.331 (0.579)
  Proliferating Cell Nuclear Antigen (PCNA) | 0.049 (0.321)
  Protein Tyrosine Phosphatase PTP-U2 (PTPRO) | -0.103 (0.691)
  C17orf87 (SCIMP) | -0.143 (0.349)
  Serpin Family G Member 1 (SERPING1) | -0.111 (0.931)
  CD353 Antigen (SLAMF8) | -0.394 (0.381)
  Stathmin 1 (STMN1) | -0.014 (0.188)
  Thyroglobulin (TG) | 0.792 (0.637)
  TIFA Inhibitor (TIFAB) | -0.120 (0.430)
  Transmembrane Protein 150B (TMEM150B) | -0.073 (0.564)
  Lymphocyte Activation Antigen CD30 (TNFRSF8) | -0.447 (0.380)
  B-Cell-Activating Factor (TNFSF13B) | -0.119 (0.346)
  Tuftelin 1 (TUFT1) | 0.279 (0.725)
  Nemitin (WDR47) | 0.117 (0.257)
  X-C Motif Chemokine Ligand 2 (XCL2) | -0.051 (0.538)

20. Secondary Outcome: Change From Baseline in Bromodomain and Extra-Terminal Domain (BET) Protein Target Gene Expression at Predose on Day 8 of Cycle 1 (21-day Cycle)
Description: Fold change from baseline (predose on Day 1 of Cycle 1 [21-day cycle]) in normalized gene expression ratios (nGER) for 49 target genes was measured to assess target engagement of BET proteins predose on Day 1 and predose on Day 8 of Cycle 1 (21-day cycle) using quantitative polymerase chain reaction (qPCR). Data were normalized by the delta-delta cycle threshold (Ct) method using housekeeping genes. Fold change from baseline was calculated as nGER at predose Day 8/baseline in logarithmic scale with a base of 2 (Log2 scale). Per protocol, target genes were assessed across all study participants by dose and this assessment was not related to any specific disease cohort. The fold change in nGER for each target gene is presented for participants pooled from the AML and DLBCL cohorts since both cohorts received the same dose. A two-fold increase in gene expression indicated a +1 Log2 fold change. Conversely, a two-fold decrease in gene expression indicated a -1 Log2 fold change.
Time Frame: Baseline (predose on Day 1 of Cycle 1) and predose on Day 8 of Cycle 1 (21-day cycle)
Population: The analysis population consisted of the total number of participants pooled from both cohorts (AML and DLBCL) who received 14 doses of MK-8628 20 mg by Day 8 of Cycle 1 (21-day cycle) and had data available for the gene expression analysis.
Measure: Mean (Standard Deviation); unit: Log2 scale fold change
Arm/Group | MK-8628 20 mg AML+DLBCL Cohorts
Number analyzed (Participants) | 8
Log2 scale fold change
  Agmatinase (AGMAT) | -0.759 (0.633)
  Annexin A3 (ANXA3) | 0.210 (0.917)
  Atonal BHLH Transcription Factor 8 (ATOH8) | -0.869 (1.059)
  B-cell Lymphoma Extra Large (BCL.xL) | 0.329 (1.964)
  B-cell Lymphoma 2 (BCL2) | -0.056 (0.450)
  Bone Marrow X-linked Kinase (BMX) | 0.115 (0.628)
  Caspase Recruitment Domain Family Member 6 (CARD6) | -0.115 (0.380)
  C-C Motif Chemokine Receptor 1 (CCR1) | -0.490 (1.185)
  Cluster of Differentiation 163 (CD163) | -0.442 (0.779)
  Choline Kinase Alpha (CHKA) | 0.218 (0.267)
  Chemerin Chemokine-Like Receptor 1 (CMKLR1) | -0.708 (1.271)
  Cysteine/Serine-Rich Nuclear Protein 2 (CSRNP2) | 0.119 (0.265)
  Dicarbonyl and L-xylulose Reductase (DCXR) | 0.696 (0.397)
  Deoxyribonuclease 1 Like 3 (DNASE1L3) | -0.386 (0.705)
  Fc Gamma Receptor Ia (FCGR1A) | -0.885 (0.348)
  Fibroblast Growth Factor Receptor 1 (FGFR1) | -0.561 (1.033)
  G Protein-Coupled Receptor 141 (GPR141) | -0.333 (1.207)
  Granzyme A (GZMA) | -0.572 (0.752)
  Granzyme B (GZMB) | -0.442 (1.402)
  Granzyme K (GZMK) | -0.657 (0.974)
  H2A Histone Family Member X (H2AFX) | 0.060 (0.466)
  Hepatitis A Virus Cellular Receptor 2 (HAVCR2) | -0.722 (0.598)
  Class B Basic Helix-Loop-Helix Protein 41 (HES6) | 0.364 (1.373)
  Hexamethylene Bisacetamide Inducible 1 (HEXIM1) | 0.429 (0.422)
  Hepatocyte Growth Factor (HGF) | -0.276 (0.383)
  Histone Cluster 2 H2B Family Member F (HIST2H2BF) | 0.427 (0.415)
  Inhibitor of Nuclear Factor-kB (IKBKE) | -0.166 (0.480)
  Interleukin 12 Receptor Subunit Beta 2 (IL12RB2) | -0.435 (1.351)
  Interleukin 7 Receptor (IL7R) | -0.301 (0.986)
  Lunatic Fringe (Drosophila) Homolog (LFNG) | 0.099 (0.668)
  Leukocyte Immunoglobulin Like Receptor A4 (LILRA4) | 0.104 (1.241)
  Macrophage Receptor (MARCO) | -1.197 (0.832)
  Membrane Spanning 4-Domains A2 (MS4A2) | 0.023 (1.266)
  Class E Basic Helix-Loop-Helix Protein 39 (MYC) | -0.270 (0.521)
  Nudix Hydrolase 12 (NUDT12) | -0.025 (0.697)
  Proliferating Cell Nuclear Antigen (PCNA) | 0.015 (0.572)
  Protein Tyrosine Phosphatase PTP-U2 (PTPRO) | -1.007 (0.839)
  C17orf87 (SCIMP) | -0.360 (1.005)
  Serpin Family G Member 1 (SERPING1) | -0.170 (1.191)
  CD353 Antigen (SLAMF8) | -0.918 (1.057)
  Stathmin 1 (STMN1) | -0.251 (0.822)
  Thyroglobulin (TG) | 0.399 (0.884)
  TIFA Inhibitor (TIFAB) | -0.937 (0.444)
  Transmembrane Protein 150B (TMEM150B) | -0.222 (0.280)
  Lymphocyte Activation Antigen CD30 (TNFRSF8) | -0.464 (0.453)
  B-Cell-Activating Factor (TNFSF13B) | -0.094 (0.445)
  Tuftelin 1 (TUFT1) | 0.472 (0.798)
  Nemitin (WDR47) | 0.263 (0.155)
  X-C Motif Chemokine Ligand 2 (XCL2) | -0.666 (0.835)

ADVERSE EVENTS:
Time Frame: Up to approximately 61 months
Description: The safety population consisted of all participants that received at least one dose of study treatment.
  The All-Cause Mortality population consisted of all randomized participants.
Arm/Group | MK-8628 20 mg AML Cohort | MK-8628 20 mg DLBCL Cohort
All-Cause Mortality (participants affected / at risk) | 3/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 20 mg AML Cohort (N=3) | MK-8628 20 mg DLBCL Cohort (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary mycosis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8628 20 mg AML Cohort (N=3) | MK-8628 20 mg DLBCL Cohort (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (6)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Factor VII deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Infusion site erythema (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 2 (2) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (3) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to limited pharmacokinetics sampling for t1/2, caution must be exercised when interpreting the results of t1/2, CL/F, and AUC 0-∞ results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT02698189/Prot_SAP_000.pdf